CLINICAL TRIAL: NCT06580704
Title: Lumbosacral Erector Spinae Plane Block Versus Psoas Muscle Compartment With Sciatic Nerve Block for Anesthesia for Unilateral Lower Limb Operations in Critically Ill Patients: A Randomized Clinical Study
Brief Title: Lumbosacral Erector Spinae Plane Block Versus Psoas Muscle Compartment With Sciatic Nerve Block for Anesthesia for Unilateral Lower Limb Operations in Critically Ill Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohammed Said ElSharkawy, Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 36264PR761/7/24
Record Dates: First submitted 2024-08-24; First posted 2024-08-30 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Lumbosacral; Erector Spinae Plane Block; Psoas Muscle Compartment Block; Sciatic Nerve Block; Anesthesia; Unilateral; Lower Limb; Critically Ill Patients

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lumbosacral Erector Spinae Plane Block (Experimental): Patients will receive ultrasound-guided lumbosacral erector spinae plane block.
  Interventions: Drug: Lumbosacral Erector Spinae Plane Block
- Psoas Muscle Compartment With Sciatic Nerve Block (Experimental): Patients will receive ultrasound-guided psoas muscle compartment with sciatic nerve block.
  Interventions: Drug: Psoas Muscle Compartment With Sciatic Nerve Block

INTERVENTIONS:
Drug: Lumbosacral Erector Spinae Plane Block — Patients will receive ultrasound-guided lumbosacral erector spinae plane block.
  Arms: Lumbosacral Erector Spinae Plane Block
Drug: Psoas Muscle Compartment With Sciatic Nerve Block — Patients will receive ultrasound-guided psoas muscle compartment with sciatic nerve block.
  Arms: Psoas Muscle Compartment With Sciatic Nerve Block

SUMMARY:
This study aims to compare lumbosacral erector spinae plane block and psoas muscle compartment with sciatic nerve block in unilateral lower limb operations in critically ill patients.

DETAILED DESCRIPTION:
The lower limb surgeries are associated with acute postoperative pain and require long-term analgesia. Regional anesthesia is often used to prevent postoperative pain. Ultrasound-guided regional anesthetic approaches provide a simple intraoperative pathway that lowers pain scores with less impact on the respiratory or cardiovascular system.

Psoas compartment block (PCB) is a peripheral regional technique of anesthesia, which provides a block of the main components of the lumbar plexus - the femoral, lateral cutaneous nerve of the femur and sciatic nerve. In combination with the sciatic nerve block, the psoas compartment block provides effective anesthesia of the entire lower extremity, with better hemodynamic stability.

The erector Spinae plane block (ESPB) is a novel regional block technique primarily introduced in 2016 for managing severe neuropathic pain.

ELIGIBILITY:
* Age from 18 to 65 years.
* Both sexes.
* American Society of Anesthesiology (ASA) physical status III, IV.
* Critically ill patients admitted to intensive care unit.
* Undergoing unilateral lower limb operations.

Exclusion Criteria:

* History of allergy to local anesthetics.
* Bleeding tendency.
* Coagulopathy.
* Anticoagulant therapy.
* Pre-existing psychological, neurologic, and spinal cord diseases.
* Previous back surgery.
* Infection or mass at the site of the block.
* Chronic analgesic therapy.
* Severe cardiac or renal diseases.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2024-08-31 (Actual); Primary Completion 2025-03-26 (Actual); Study Completion 2025-03-26 (Actual)

PRIMARY OUTCOMES:
Incidence of failure | Intraoperatively
  Incidence of failure will be recorded. After 30minutes, the pinprick test will be performed. If pain persists, the patient will be excluded.

SECONDARY OUTCOMES:
Hear rate | Every 15 minutes till the end of surgery (up to 2 hours)
  Hear rate will be recorded preoperative, before performing of block, and every 15 minutes till the end of surgery.
Mean arterial pressure | Every 15 minutes till the end of surgery (up to 2 hours)
  Mean arterial pressure will be recorded preoperative, before performing of block, and every 15 minutes till the end of surgery.
Duration of analgesia | Till the first request of rescue analgesic drug (up to 24 hours after surgery)
  Duration of analgesia (time from the injection of anesthetic solution to the first request of rescue analgesic drug) will be assessed.
Degree of pain | 24 hours postoperatively
  Each patient will be instructed about postoperative pain assessment with the visual analogue scale (VAS). VAS (0 represents "no pain" while 10 represents "the worst pain imaginable"). VAS will be assessed at PACU, 2, 4, 6, 8, 12, and 24 h postoperatively.
Degree of patient satisfaction | 24 hours postoperatively
  The degree of patient satisfaction will be assessed on a 5-point Likert scale patient satisfaction (1, extremely dissatisfied; 2, unsatisfied; 3, neutral; 4, satisfied; 5, extremely satisfied).
Incidence of adverse events | 24 hours postoperatively
  Incidence of adverse events such as local anesthetic systemic toxicity (LAST), bradycardia, hypotension, postoperative nausea and vomiting (PONV), hematoma, or any other complication will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.